CLINICAL TRIAL: NCT02598271
Title: Influence of Elevated Baseline Serum Creatinine and Body Composition on Acute Kidney Injury in Cardiac Surgery - The InCreAS Trial
Brief Title: Influence of Elevated Baseline Serum Creatinine and Body Composition on Acute Kidney Injury in Cardiac Surgery
Acronym: InCreAS
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Martin Bernardi, Dr., Medical University of Vienna
Other Study IDs: 1223/2015
Record Dates: First submitted 2015-11-01; First posted 2015-11-05 (Estimated); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Acute Kidney Injury
Keywords: Acute Kidney Injury; Cardiac Surgery
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Low SCr: Patients with a serum creatinine below or equal to 1.3mg/dL
- High SCr: Patients with a serum creatinine above to 1.3mg/dL

SUMMARY:
Acute kidney injury (AKI) is an infrequent but major and well - recognized complication of cardiac surgery. Recent studies demonstrated that even minimal increases in serum creatinine are associated with a rising risk of mortality, hospital length of stay, and cost. Furthermore a cut-off for baseline serum creatinine and its influence on mortality after cardiac surgery has been shown.

In this study the investigators want to test if increased bSCr is influenced by body composition. Further the investigators want to determine if the incidence of AKI is different in patients below or above the estimated cut-off. Therefore the investigators want to perform a prospective cohort analysis and will take several other body composition and nutrition parameters to test their influence on the predictive power of bSCr. Furthermore the investigators want to evaluate several novel biomarkers for AKI on their predictive effect in cardiac surgical patients.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is an infrequent but major and well - recognized complication of cardiac surgery (1, 2). Its incidence ranges from 1 to 30% (3). Numerous pre-, intra-, and postoperative factors have been associated with the development of AKI after cardiac surgery (3-19). Most commonly used definitions are the absolute serum creatinine level, its change within one week and/or the need for dialysis in previously undialysed patients (1, 3-5, 9-11, 19-25). In patients who are older, more obese with Type 2 diabetes and hypertension, there is increasing interest in the effects of chronic kidney disease on the cardiovascular system (26). Recent studies demonstrated that even minimal increases in serum creatinine are associated with a rising risk of mortality, hospital length of stay, and cost (27, 28). The Acute Dialysis Quality Initiative Group standardized with their Risk, Injury, Failure, Loss of Kidney Function, End-Stage Kidney Disease criteria and their modifications to the Acute Kidney Injury Network criteria the definitions of AKI (19, 29, 30). Both criteria need a baseline serum creatinine value for estimation (31).

In a recent published study (32) a cut-off for baseline serum creatinine and its influence on mortality after cardiac surgery has been shown. Under the steady-state and stable kidney function, SCr is usually produced at a relatively constant rate by the body depending on the absolute amount of muscle mass, and is a reliable and cost-effective surrogate marker for kidney function (33). SCr is strongly correlated with weight, total body water and anthropometrically estimated lean body mass (LBM) (34). Approximately half of LBM is comprised of skeletal muscle mass (35). Recent studies suggest that higher muscle mass is associated with greater longevity in people with CKD and other chronic disease states (36, 37). SCr, however, has several limitations, such as variations in concentration related to age, sex, muscle mass and is influenced by dietary protein intake. (38) Furthermore AKI affects different complex cellular and molecular pathways. Several novel urinary biomarkers such as insulin-like growth factor-binding protein 7 (IGFBP7), tissue inhibitor of metalloproteinases-2 (TIMP-2) and neutral endopeptidase (NEP) are involved in the early phase of cell injury and predict both the development and severity of AKI and renal recovery early after cardiac surgery (39-43) In this study the investigators want to test if increased bSCr is influenced by body composition. Further the investigators want to determine if the incidence of AKI is different in patients below or above the estimated cut-off. Therefore the investigators want to perform a prospective cohort analysis and will take several other body composition and nutrition parameters to test their influence on the predictive power of bSCr. Furthermore the investigators want to evaluate several novel biomarkers for AKI on their predictive effect in cardiac surgical patients.

ELIGIBILITY:
Inclusion Criteria:

* Elective cardiac surgical intervention

Exclusion Criteria:

* Emergency procedures
* Heart transplantation
* Elective left ventricular assist device (LVAD) implantation o Pulmonary thrombendarterectomy
* Declined informed consent
* Age < 18 years
* Pregnant woman
* Preoperative renal replacement therapy (RRT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing an elective cardiac surgical intervention.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-08-12 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Influence of body composition on increased baseline serum creatinine | 7 days
  Body composition will be measured by bioelectrical impedance analysis, body weight, muscle status and nutrition status

SECONDARY OUTCOMES:
Influence of increased baseline serum creatinine on difference in acute kidney injury after cardiac surgery | 7 days
  Acute kidney injury will be defined by current KDIGO-Guidelines for acute kidney inujury
Influence of neutral endopeptidase on levels of acute kidney injury | 7 days
  Neutral endopeptidase will be measured out of the urine with ELISA
Influence of right ventricular function on acute kidney injury | 7 days
  Right ventricular function will be assessed by Tricuspid annular plane systolic excursion (TAPSE) measurements
Length of ICU stay | 7 days
30 days mortality | 30 days
Volume status | 7 days
  Need of crystalloid, colloid and blood products
Influence of podocin on levels of acute kidney injury | 7 days
  Podocin will be measured out of the urine with ELISA
Influence of nephrin on levels of acute kidney injury | 7 days
  Nephrin will be measured out of the urine with ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Martin H Bernardi, Dr., Principal Investigator — Divison of Cardiothoracic Anaesthesia and Intensive Care, Medical University of Vienna
Locations (1):
- Divison of Cardiothoracic Anaesthesia and Intensive Care, Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Background] Ostermann ME, Taube D, Morgan CJ, Evans TW. Acute renal failure following cardiopulmonary bypass: a changing picture. Intensive Care Med. 2000 May;26(5):565-71. doi: 10.1007/s001340051205. PMID 10923731
- [Background] Chertow GM, Levy EM, Hammermeister KE, Grover F, Daley J. Independent association between acute renal failure and mortality following cardiac surgery. Am J Med. 1998 Apr;104(4):343-8. doi: 10.1016/s0002-9343(98)00058-8. PMID 9576407
- [Background] Mangano CM, Diamondstone LS, Ramsay JG, Aggarwal A, Herskowitz A, Mangano DT. Renal dysfunction after myocardial revascularization: risk factors, adverse outcomes, and hospital resource utilization. The Multicenter Study of Perioperative Ischemia Research Group. Ann Intern Med. 1998 Feb 1;128(3):194-203. doi: 10.7326/0003-4819-128-3-199802010-00005. PMID 9454527
- [Background] Bahar I, Akgul A, Ozatik MA, Vural KM, Demirbag AE, Boran M, Tasdemir O. Acute renal failure following open heart surgery: risk factors and prognosis. Perfusion. 2005 Oct;20(6):317-22. doi: 10.1191/0267659105pf829oa. PMID 16363316
- [Background] Janssen DP, Noyez L, van Druten JA, Skotnicki SH, Lacquet LK. Predictors of nephrological morbidity after coronary artery bypass surgery. Cardiovasc Surg. 2002 Jun;10(3):222-7. doi: 10.1016/s0967-2109(01)00134-x. PMID 12044429
- [Background] Aronson S, Boisvert D, Lapp W. Isolated systolic hypertension is associated with adverse outcomes from coronary artery bypass grafting surgery. Anesth Analg. 2002 May;94(5):1079-84, table of contents. doi: 10.1097/00000539-200205000-00005. PMID 11973166
- [Background] Aronson S, Fontes ML, Miao Y, Mangano DT; Investigators of the Multicenter Study of Perioperative Ischemia Research Group; Ischemia Research and Education Foundation. Risk index for perioperative renal dysfunction/failure: critical dependence on pulse pressure hypertension. Circulation. 2007 Feb 13;115(6):733-42. doi: 10.1161/CIRCULATIONAHA.106.623538. Epub 2007 Feb 5. PMID 17283267
- [Background] Mangano DT, Tudor IC, Dietzel C; Multicenter Study of Perioperative Ischemia Research Group; Ischemia Research and Education Foundation. The risk associated with aprotinin in cardiac surgery. N Engl J Med. 2006 Jan 26;354(4):353-65. doi: 10.1056/NEJMoa051379. PMID 16436767
- [Background] Gaudino M, Luciani N, Giungi S, Caradonna E, Nasso G, Schiavello R, Luciani G, Possati G. Different profiles of patients who require dialysis after cardiac surgery. Ann Thorac Surg. 2005 Mar;79(3):825-9; author reply 829-30. doi: 10.1016/j.athoracsur.2004.08.019. PMID 15734386
- [Background] Kincaid EH, Ashburn DA, Hoyle JR, Reichert MG, Hammon JW, Kon ND. Does the combination of aprotinin and angiotensin-converting enzyme inhibitor cause renal failure after cardiac surgery? Ann Thorac Surg. 2005 Oct;80(4):1388-93; discussion 1393. doi: 10.1016/j.athoracsur.2005.03.136. PMID 16181876
- [Background] Regner KR, Connolly HM, Schaff HV, Albright RC. Acute renal failure after cardiac surgery for carcinoid heart disease: incidence, risk factors, and prognosis. Am J Kidney Dis. 2005 May;45(5):826-32. doi: 10.1053/j.ajkd.2005.02.009. PMID 15861347
- [Background] Mehta RH, Bruckman D, Das S, Tsai T, Russman P, Karavite D, Monaghan H, Sonnad S, Shea MJ, Eagle KA, Deeb GM. Implications of increased left ventricular mass index on in-hospital outcomes in patients undergoing aortic valve surgery. J Thorac Cardiovasc Surg. 2001 Nov;122(5):919-28. doi: 10.1067/mtc.2001.116558. PMID 11689797
- [Background] Fischer UM, Weissenberger WK, Warters RD, Geissler HJ, Allen SJ, Mehlhorn U. Impact of cardiopulmonary bypass management on postcardiac surgery renal function. Perfusion. 2002 Nov;17(6):401-6. doi: 10.1191/0267659102pf610oa. PMID 12470028
- [Background] Aronson S, Dyke CM, Stierer KA, Levy JH, Cheung AT, Lumb PD, Kereiakes DJ, Newman MF. The ECLIPSE trials: comparative studies of clevidipine to nitroglycerin, sodium nitroprusside, and nicardipine for acute hypertension treatment in cardiac surgery patients. Anesth Analg. 2008 Oct;107(4):1110-21. doi: 10.1213/ane.0b013e31818240db. PMID 18806012
- [Background] Brown JR, Cochran RP, Leavitt BJ, Dacey LJ, Ross CS, MacKenzie TA, Kunzelman KS, Kramer RS, Hernandez F Jr, Helm RE, Westbrook BM, Dunton RF, Malenka DJ, O'Connor GT; Northern New England Cardiovascular Disease Study Group. Multivariable prediction of renal insufficiency developing after cardiac surgery. Circulation. 2007 Sep 11;116(11 Suppl):I139-43. doi: 10.1161/CIRCULATIONAHA.106.677070. PMID 17846294
- [Background] Arora P, Rajagopalam S, Ranjan R, Kolli H, Singh M, Venuto R, Lohr J. Preoperative use of angiotensin-converting enzyme inhibitors/angiotensin receptor blockers is associated with increased risk for acute kidney injury after cardiovascular surgery. Clin J Am Soc Nephrol. 2008 Sep;3(5):1266-73. doi: 10.2215/CJN.05271107. Epub 2008 Jul 30. PMID 18667735
- [Background] Maslow AD, Chaudrey A, Bert A, Schwartz C, Singh A. Perioperative renal outcome in cardiac surgical patients with preoperative renal dysfunction: aprotinin versus epsilon aminocaproic acid. J Cardiothorac Vasc Anesth. 2008 Feb;22(1):6-15. doi: 10.1053/j.jvca.2007.07.017. Epub 2007 Nov 7. PMID 18249324
- [Background] Salis S, Mazzanti VV, Merli G, Salvi L, Tedesco CC, Veglia F, Sisillo E. Cardiopulmonary bypass duration is an independent predictor of morbidity and mortality after cardiac surgery. J Cardiothorac Vasc Anesth. 2008 Dec;22(6):814-22. doi: 10.1053/j.jvca.2008.08.004. Epub 2008 Oct 22. PMID 18948034
- [Background] Weir MR, Aronson S, Avery EG, Pollack CV Jr. Acute kidney injury following cardiac surgery: role of perioperative blood pressure control. Am J Nephrol. 2011;33(5):438-52. doi: 10.1159/000327601. Epub 2011 Apr 21. PMID 21508632
- [Background] Swaminathan M, Shaw AD, Phillips-Bute BG, McGugan-Clark PL, Archer LE, Talbert S, Milano CA, Patel UD, Stafford-Smith M. Trends in acute renal failure associated with coronary artery bypass graft surgery in the United States. Crit Care Med. 2007 Oct;35(10):2286-91. doi: 10.1097/01.ccm.0000282079.05994.57. PMID 17944016
- [Background] Bove T, Calabro MG, Landoni G, Aletti G, Marino G, Crescenzi G, Rosica C, Zangrillo A. The incidence and risk of acute renal failure after cardiac surgery. J Cardiothorac Vasc Anesth. 2004 Aug;18(4):442-5. doi: 10.1053/j.jvca.2004.05.021. PMID 15365924
- [Background] Chertow GM, Lazarus JM, Paganini EP, Allgren RL, Lafayette RA, Sayegh MH. Predictors of mortality and the provision of dialysis in patients with acute tubular necrosis. The Auriculin Anaritide Acute Renal Failure Study Group. J Am Soc Nephrol. 1998 Apr;9(4):692-8. doi: 10.1681/ASN.V94692. PMID 9555672
- [Background] Leacche M, Rawn JD, Mihaljevic T, Lin J, Karavas AN, Paul S, Byrne JG. Outcomes in patients with normal serum creatinine and with artificial renal support for acute renal failure developing after coronary artery bypass grafting. Am J Cardiol. 2004 Feb 1;93(3):353-6. doi: 10.1016/j.amjcard.2003.10.020. PMID 14759390
- [Background] Thakar CV, Worley S, Arrigain S, Yared JP, Paganini EP. Influence of renal dysfunction on mortality after cardiac surgery: modifying effect of preoperative renal function. Kidney Int. 2005 Mar;67(3):1112-9. doi: 10.1111/j.1523-1755.2005.00177.x. PMID 15698452
- [Background] Doddakula K, Al-Sarraf N, Gately K, Hughes A, Tolan M, Young V, McGovern E. Predictors of acute renal failure requiring renal replacement therapy post cardiac surgery in patients with preoperatively normal renal function. Interact Cardiovasc Thorac Surg. 2007 Jun;6(3):314-8. doi: 10.1510/icvts.2006.148874. Epub 2007 Mar 7. PMID 17669854
- [Background] McCullough PA, Haapio M, Mankad S, Zamperetti N, Massie B, Bellomo R, Berl T, Anker SD, Anand I, Aspromonte N, Bagshaw SM, Bobek I, Cruz DN, Daliento L, Davenport A, Hillege H, House AA, Katz N, Maisel A, Mebazaa A, Palazzuoli A, Ponikowski P, Ronco F, Shaw A, Sheinfeld G, Soni S, Vescovo G, Zanco P, Ronco C, Berl T; Acute Dialysis Quality Initiative (ADQI) Consensus Group. Prevention of cardio-renal syndromes: workgroup statements from the 7th ADQI Consensus Conference. Nephrol Dial Transplant. 2010 Jun;25(6):1777-84. doi: 10.1093/ndt/gfq180. Epub 2010 Apr 6. No abstract available. PMID 20375030
- [Background] Chertow GM, Burdick E, Honour M, Bonventre JV, Bates DW. Acute kidney injury, mortality, length of stay, and costs in hospitalized patients. J Am Soc Nephrol. 2005 Nov;16(11):3365-70. doi: 10.1681/ASN.2004090740. Epub 2005 Sep 21. PMID 16177006
- [Background] Lassnigg A, Schmidlin D, Mouhieddine M, Bachmann LM, Druml W, Bauer P, Hiesmayr M. Minimal changes of serum creatinine predict prognosis in patients after cardiothoracic surgery: a prospective cohort study. J Am Soc Nephrol. 2004 Jun;15(6):1597-605. doi: 10.1097/01.asn.0000130340.93930.dd. PMID 15153571
- [Background] Srisawat N, Hoste EE, Kellum JA. Modern classification of acute kidney injury. Blood Purif. 2010;29(3):300-7. doi: 10.1159/000280099. Epub 2010 Feb 3. PMID 20130395
- [Background] Bellomo R, Ronco C, Kellum JA, Mehta RL, Palevsky P; Acute Dialysis Quality Initiative workgroup. Acute renal failure - definition, outcome measures, animal models, fluid therapy and information technology needs: the Second International Consensus Conference of the Acute Dialysis Quality Initiative (ADQI) Group. Crit Care. 2004 Aug;8(4):R204-12. doi: 10.1186/cc2872. Epub 2004 May 24. PMID 15312219
- [Background] Zavada J, Hoste E, Cartin-Ceba R, Calzavacca P, Gajic O, Clermont G, Bellomo R, Kellum JA; AKI6 investigators. A comparison of three methods to estimate baseline creatinine for RIFLE classification. Nephrol Dial Transplant. 2010 Dec;25(12):3911-8. doi: 10.1093/ndt/gfp766. Epub 2010 Jan 25. PMID 20100732
- [Background] Bernardi MH, Schmidlin D, Schiferer A, Ristl R, Neugebauer T, Hiesmayr M, Druml W, Lassnigg A. Impact of preoperative serum creatinine on short- and long-term mortality after cardiac surgery: a cohort study. Br J Anaesth. 2015 Jan;114(1):53-62. doi: 10.1093/bja/aeu316. Epub 2014 Sep 19. PMID 25240162
- [Background] Heymsfield SB, Arteaga C, McManus C, Smith J, Moffitt S. Measurement of muscle mass in humans: validity of the 24-hour urinary creatinine method. Am J Clin Nutr. 1983 Mar;37(3):478-94. doi: 10.1093/ajcn/37.3.478. PMID 6829490
- [Background] Schutte JE, Longhurst JC, Gaffney FA, Bastian BC, Blomqvist CG. Total plasma creatinine: an accurate measure of total striated muscle mass. J Appl Physiol Respir Environ Exerc Physiol. 1981 Sep;51(3):762-6. doi: 10.1152/jappl.1981.51.3.762. PMID 7327978
- [Background] Lee RC, Wang Z, Heo M, Ross R, Janssen I, Heymsfield SB. Total-body skeletal muscle mass: development and cross-validation of anthropometric prediction models. Am J Clin Nutr. 2000 Sep;72(3):796-803. doi: 10.1093/ajcn/72.3.796. PMID 10966902
- [Background] von Herrath M, Holzer H. Oxidative inactivation of yeast fructose-1,6-bisphosphatase. Prog Clin Biol Res. 1985;180:329-40. PMID 2994088
- [Background] Solntseva EI, Borisova OV. [Imidazole causes long-term elevation of evoked postsynaptic potential and potential-dependent calcium current in molluskan neurons]. Dokl Akad Nauk SSSR. 1988;300(3):760-3. No abstract available. Russian. PMID 2844485
- [Background] Patel SS, Molnar MZ, Tayek JA, Ix JH, Noori N, Benner D, Heymsfield S, Kopple JD, Kovesdy CP, Kalantar-Zadeh K. Serum creatinine as a marker of muscle mass in chronic kidney disease: results of a cross-sectional study and review of literature. J Cachexia Sarcopenia Muscle. 2013 Mar;4(1):19-29. doi: 10.1007/s13539-012-0079-1. Epub 2012 Jul 10. PMID 22777757
- [Background] Devarajan P. Update on mechanisms of ischemic acute kidney injury. J Am Soc Nephrol. 2006 Jun;17(6):1503-20. doi: 10.1681/ASN.2006010017. Epub 2006 May 17. No abstract available. PMID 16707563
- [Background] Rodier F, Campisi J, Bhaumik D. Two faces of p53: aging and tumor suppression. Nucleic Acids Res. 2007;35(22):7475-84. doi: 10.1093/nar/gkm744. Epub 2007 Oct 16. PMID 17942417
- [Background] Boonstra J, Post JA. Molecular events associated with reactive oxygen species and cell cycle progression in mammalian cells. Gene. 2004 Aug 4;337:1-13. doi: 10.1016/j.gene.2004.04.032. PMID 15276197
- [Background] Meersch M, Schmidt C, Van Aken H, Martens S, Rossaint J, Singbartl K, Gorlich D, Kellum JA, Zarbock A. Urinary TIMP-2 and IGFBP7 as early biomarkers of acute kidney injury and renal recovery following cardiac surgery. PLoS One. 2014 Mar 27;9(3):e93460. doi: 10.1371/journal.pone.0093460. eCollection 2014. PMID 24675717
- [Background] Truong LD, Shen SS. Immunohistochemical diagnosis of renal neoplasms. Arch Pathol Lab Med. 2011 Jan;135(1):92-109. doi: 10.5858/2010-0478-RAR.1. PMID 21204715